CLINICAL TRIAL: NCT05495412
Title: A Single Case Study to Explore the Impact of Community-based Rebound Therapy on Chest Health Outcomes in School Aged Children and Young People With Neurodisability and Respiratory Issues.
Brief Title: Rebound for Respiratory in School Aged Children and Young People With Neurodisability
Acronym: RforR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jon Marsden (Other)
Collaborators: UCL Great Ormond Street Institute of Child Health (Other)
Responsible Party: Sponsor-Investigator, Jon Marsden, Professor of Rehabilitation, University of Plymouth
Organization: University of Plymouth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2698; NIHR301008 (Other Grant/Funding Number: National Institute of Health Research)
Record Dates: First submitted 2022-04-28; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Disorder; Respiratory Tract Infections
MeSH Terms: conditions — Nervous System Diseases; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: single case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rebound therapy (Other): Exercise therapy which uses a full sized trampoline to provide opportunities for movement, therapeutic exercise and recreation for children and young people.
  Interventions: Other: Rebound therapy

INTERVENTIONS:
Other: Rebound therapy — Exercise therapy delivered twice weekly for 6 weeks, during Phase B of an ABA single case study design.

SUMMARY:
Background:

Respiratory illness is the most common reason to attend primary and hospital care in children with neurodisability, accruing significant healthcare costs. Moreover, it remains the primary cause of death in this population. Exercise plays an important role in the prevention and management of respiratory illness in children with neurodisability. Rebound therapy is a popular form of therapeutic exercise using trampolines to facilitate movement. It is highly accessible for children with complex neurodisabilities and has been shown to improve muscle tone, balance, sitting posture, behaviour and quality of life. Additional chest health benefits have been observed in other populations, but has yet to be established in children with neurodisability.

Aim:

This clinical study seeks to explore the impact of community-based rebound therapy on chest health outcomes in school-aged children and young people with complex neurodisability and respiratory issues.

Method:

A single case study ABA design, inviting 4-6 children with neurodisability and respiratory issues to participate. The study will comprise of:

Phase A: 6-week observational baseline measures alongside usual care Phase B: 6-week of rebound therapy, delivered twice weekly alongside usual care Phase A: 6-week observational follow up measures alongside usual care.

Measurements:

1. Chest health parameters, measured using respiratory rate, cough frequency, time taken to complete chest care, hospital days, emergency days and primary care consultation days
2. Caregiver-reported chest health, measured using the Respiratory Questionnaire for Children with Neurological Impairment questionnaire.
3. Caregiver reported quality of life, measured using the CPCHILD Questionnaire and an optional exit interview at week 18 of the study
4. Posture will be measured using the Chailey Levels of Ability Scale.
5. Adverse Events, measured through safety monitoring of new symptoms, worsening symptoms, hospital days, emergency department days and primary consultation days.
6. Adherence, measured through % attendance to 12 rebound sessions.

Data Analysis:

For each single case study, serial data will be subjected to within-phase (A) analysis of stability criterion and across phase (AB) analysis. Single outcome measure data will be plotted alongside serial data findings, providing visual analysis and interpretation of trends. The exit interview will provide textual data that will be subject to thematic analysis methods.

Anticipated Results:

Results will provide early proof of concept data informing the short term effects of exercise-based rebound therapy intervention on chest health, posture and quality of life for children with complex neurodisabilities.

A composite of passive respiratory clinical measurements and participant/caregiver-reported outcomes will be proposed, implementing a combination of serial and single measurements to inform feasibility of future hypothesis testing research.

The close monitoring of adverse events and adherence will inform safety of intervention prescribed and feasibility of delivering intervention to children with complex neurodisabilities and respiratory impairment.

DETAILED DESCRIPTION:
This study protocol seeks to explore the impact of community-based rebound therapy on chest health outcomes in school-aged children and young people with complex neurodisability and respiratory issues.

Neurodisability represents one of the largest populations of childhood disability in the UK, defined as a group of conditions associated with impairment of the nervous system. Within this population, respiratory illness is the most common reason to attend primary care consultation, emergency hospital admission and intensive care, accruing significant healthcare costs. Moreover, it remains the primary cause of death, accounting for 51% of cases in children with cerebral palsy.

Chronic respiratory impairments within paediatric neurodisability demand long-term management beyond acute transitory exacerbation, directing attention to prevention and community-based management of respiratory disease. A recent consensus study highlights the importance of optimising physical activity and fitness, postural management and airway clearance in this population, although evidence is limited by lack of comparison groups and good outcome measures. A recent Cochrane review identifies a wide diversity of anecdotally beneficial treatments to support respiratory health within this population of interest, but recognises no 'gold standard' non-pharmaceutical intervention consensus, limited by few and poor-quality studies. However, this body of available literature offers hypothesis generating findings, informing a wide scope for future research into preventing and managing respiratory impairment in children with neurodisability.

Exercise has been identified as a key intervention in the prevention and management of respiratory disease in children with neurodisability. Rebound therapy is a popular form of exercise established in UK educational settings and uses trampolines to provide highly accessible therapeutic exercise to children with moderate to severe complex needs where participation in exercise is otherwise limited. Studies have found rebound therapy to improve participation, muscle tone, and balance, sitting position, behaviour and quality of life in children with neurodisability and features as an important component of care standards for people with learning disability.

Additional respiratory benefits of rebound therapy have also been established in children with cystic fibrosis. Yet, within the population of interest, claims have not been thoroughly examined. There is some evidence to suggest rebound therapy could be advantageous for children with moderate to severe neurodisability, who cannot actively participate in airway clearance techniques and those with a weak cough. Small scale studies indicate improved lung volumes through movement, vocalisation and laughing and imitation of percussion and vibration techniques through the bounce of the trampoline. This raises hypothesis generating evidence that demands further research to establish the effects of this highly accessible, multi-beneficial form of exercise.

This study's primary aim is to explore the impact of rebound therapy on chest health in children with neurodisability and respiratory impairment.

Primary Objective

Objective 1) To explore the impact of a 6-week customised rebound therapy programme on chest health outcomes in children with neurodisability and respiratory issues. This will be primarily measured Respiratory Questionnaire For Children with Neurological Impairment.

Secondary measurements will include:

* Respiratory health recordings via text, including respiratory per minute, cough frequency per minute and time spent completing respiratory care in predetermined period of time. Oxygen saturations will be included if measured as part of an individual's usual care.
* Participant/caregiver-reported changes in general health
* Participant/caregiver-reported changes in 'usual' chest care
* Escalation of chest care: attended days for primary care consult, emergency department and/or hospital admission.

Secondary Objectives

Objective 2) To explore the impact of a 6-week customised rebound therapy programme on participant /caregiver-reported quality of life (QoL) in children with neurodisability and respiratory issues. This will be measured using:

* Caregiver-reported CPCHILD questionnaire
* Semi-structured exit interview exploring perceived views of QoL indicators. The topic guide will explore communication, emotional wellbeing, pain, mobility, self-care /independence, social activities, worry /mental health, sleep, behaviour and safety.

Objective 3) To explore the impact of a 6-week customised rebound therapy programme on postural management outcomes in children with neurodisability and respiratory issues. This will be measured using:

* Chailey Levels of Ability Scale
* Participant/caregiver-reported changes in 'usual' postural management care plan

Objective 4) To monitor adherence to a 6-week customised rebound therapy programme, with reasons for non-adherence documented. This will be measured through recording % of rebound therapy sessions attended and reason for non-attendance.

Objective 5) To monitor (S) AE's during the study period, during usual care and during the 6-week customised rebound therapy programme. This will be measured through weekly respiratory health recordings via text and participant/caregiver telephone follow up.

Exploratory Objectives

Objective 6) To explore parent/caregiver perceptions of the study design components, outcome measures and contact methods. This will be measured through the semi-structured exit interview.

Methods:

The study is a single case design, recruiting N=4-6 participants. This study design has been selected in the absence of existing published research, to examine a relationship between rebound therapy intervention and change in respiratory outcomes in CYP with neurodisability. A broad spectrum of variables will be examined, contributing both quantitative and qualitative data that offer dynamic and flexible findings unique to each single case study. However, the intervention will be examined under a given set of conditions aligning with a deductive/static approach to facilitate comparison and similarities across a heterogeneous cohort.

Each single case study will replicate an ABA design, incorporating:

* Phase A baseline measures at week 0
* Phase B pre-intervention measures at week 6
* Phase B post-intervention measures at week 12
* Phase A follow up measure at week 18. Clinical outcome measures requiring participant/caregiver clinic attendance will be conducted at the four data time points specified above. Serial outcome measurements that do not require participant/caregiver clinic attendance will be conducted at weekly intervals during the study period (week 0-18) to reduce participant travel and burden.

Study Setting:

The study will be conducted across three sites:

* A clinical NHS site accessed to undertake clinical measurements at week 0, 6, 12 and 18.
* Two clinical Non-NHS sites, based within community special education settings in Torbay and South Devon.

In the event that schools can facilitate safe access to parents/caregivers, the family will be provided with a choice to attend clinical outcome measurements in the therapy room of their educational setting as an alternative to the clinical NHS site, in an aim to reduce travel burden for the participant.

Recruitment

Potential participants and will be identified through paediatric clinicians working within Child and Family Health Devon. Those who express an interest in taking part will be sent an information pack, consisting of a consent to contact form and a participant information sheet (PIS) for parent/caregiver(s) and their child. Potential participants and/or their caregiver(s) will be asked to read the information provided and return the consent to contact form, confirming their interest in participation, likely eligibility and consent for the PI to contact them for eligibility screening.

Study procedures:

Eligibility Screening: This process will be completed with participant/caregiver(s) via telephone. If eligible, a baseline assessment will be booked within 2 weeks and verbal consent gained to post a questionnaire booklet (containing the CPCHILD and Respiratory Questionnaire For Children with Neurological Impairment), to be completed prior to baseline appointment to be completed prior to baseline appointment.

Phase A: BASELINE OBSERVATION

Week 0 Summary of face to face contact:

* Consent procedure
* Information gathering
* Chailey Levels of Ability Scale
* Completion of CPCHILD
* Completion of Respiratory Questionnaire For Children with Neurological Impairment Week 0-6 Summary of weekly remote contact
* Participant/caregiver-reported clinical parameter reporting
* Participant/caregiver-reported general, respiratory and postural management health
* Participant/caregiver-reported adverse event safety monitoring of new symptoms, worsening symptoms, hospital admission days, emergency department days, primary care consultation days.

Phase B INTERVENTION:

Week 6 (pre-intervention) Summary of face to face contact:

* Chailey Levels of Ability Scale
* Completion of CPCHILD
* Completion of Respiratory Questionnaire For Children with Neurological Impairment Week 6-12 Summary of face to face contact
* Twice weekly rebound therapy Week 6-12 Summary of weekly remote contact
* Participant/caregiver-reported clinical parameter reporting
* Participant/caregiver-reported general, respiratory and postural management health
* Participant/caregiver-reported adverse event safety monitoring of new symptoms, worsening symptoms, hospital admission days, emergency department days, primary care consultation days.

Phase A: FOLLOW UP OBSERVATION

Week 12 (post intervention) Summary of face to face contact:

* Chailey Levels of Ability Scale
* Completion of CPCHILD
* Completion of Respiratory Questionnaire For Children with Neurological Impairment

Week 12-18 Summary of weekly remote contact:

* Participant/caregiver-reported clinical parameter reporting
* Participant/caregiver-reported general, respiratory and postural management health
* Participant/caregiver-reported adverse event safety monitoring of new symptoms, worsening symptoms, hospital admission days, emergency department days, primary care consultation days.

Week 18 Summary of face to face contact:

* Chailey Levels of Ability Scale
* Completion of CPCHILD
* Completion of Respiratory Questionnaire For Children with Neurological Impairment
* Exit interview (optional)

Data Analysis Plan

Outcome analysis of serial measurements

For each single case study, serial data will be plotted on a line graph and subjected to:

* Within-phase (A) analysis of stability criterion
* Across phase (AB) analysis using an extended celeration line (ECL), a percentage of overlapping data (PND) and where within-phase stability criterion is satisfied, a Two Standard Deviation Band Method.

Outcome analysis of single measurements Data from the single outcome measures, defined as those collecting N=4 data points across the study period, such as caregiver reported chest health, posture and QoL will be plotted on a line graph for each single case study participant. The graph will provide visual analysis and interpretation of trends, which will be compared alongside findings from serial measurement data analysis.

Outcome analysis of qualitative data

For each single-case study, textual data will be subject to thematic analysis methods. This data will be obtained from two sources:

* Serial prospective data collected via participant/caregiver reported recordings via Text
* Single retrospective narratives shared during the exit interview

Text data will be compiled for each single-case study, maintaining timelines of serial textual data collected to facilitate comparison with quantitative data. Text data from the exit interview will be transcribed by the PI. All textual data will be uploaded into NVIVO 12 software programme to facilitate organisation of the coding process within each case-study and across case-studies.

Transcripts will be reviewed in-depth to develop familiarisation of the text. Data will be dissembled to create meaningful grouping. Emerging codes will be allocated to text fragments, identifying interesting features and grouping these through similarities and differences. These codes may be revised during the process of reading. For the purpose of rigour, a small sample of data will be analysed by a second person in the research team. The codes will be mapped across the case studies and conceptualised into themes. Themes may offer development of subthemes. Finally, the themes, sub-themes and representative text fragments will be presented in relation to the study objectives and triangulated with quantitative data analysis to generate understanding or context.

The exit interview will provide textual data that will be subject to thematic analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Age: >4 years up to <16years
* Access to a caregiver in a position of main custody, capable of giving consent on the participant's behalf
* Access to a caregiver in a position of main custody who is able to consent to also participate in the study
* Accesses full time education
* Clinical diagnosis of neurodisability
* Physical impairment Gross Motor Function Classification Scale level 3-5 defined as: (Level 3): Walks with aids. Uses wheelchair for long distances; (Level 4): Self mobility with powered mobility; (Level 5): Severely limited, unable to lift head and trunk or use powered mobility due to other comorbidities like vision impairment.
* Swallow impairment Eating Drinking Ability Classification Scale Level 3-5, defined as (Level 3): Eats and drinks with some limitations to safety; maybe limitations to efficiency; (Level 4): Eats and drinks with significant limitations to safety; (Level 5): Unable to eat or drink safely - tube feeding may be considered to provide nutrition
* Symptoms of respiratory impairment, experienced at least once a week, defined as one or more of the following: (1) Noisy breathing (wheezy, gurgling, rattily etc.); (2) Weak/poor cough; (3) Difficulty clearing secretions AND a history of a chest infection in the past 3 years requiring medication.
* Risk assessment of safe access to educational setting
* Risk assessment of contraindications and care factors for rebound therapy

Exclusion Criteria:

* Children diagnosed with a progressive neurological presentation, including muscular dystrophies.
* Children with a confirmed absolute contraindication that will determine the participant unsuitable to participate in rebound therapy. These include: (1)Cranio-vertebral Instability (including Atlanto-Axial Instability & Atlanto-Occipital Instability); (2) Detatching retina (s) or repaired retina (s); (3) Pregnancy; (4) Brittle bones; (5) Dwarfism; (6) Spinal rodding.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver-reported respiratory symptoms between week 0, 6, 12 and week 18 | Proposed Measurement point: week 0, 6, 12, and 18.
  Self/proxy reported respiratory symptoms in the last month, using the Respiratory Questionnaire For Children with Neurological Impairment

SECONDARY OUTCOMES:
Change in Clinical Respiratory Observations | Proposed Measurement points: serial weekly measurements from week 0-18.
  Self/proxy reported respiratory symptoms Participant/caregivers will be asked to report on respiratory health recordings via text (RR per minute, cough frequency per minute, time spent completing respiratory care in predetermined period of time). Oxygen saturations will be included only if a saturation monitor is available as part of an individual's usual care.
Change in Chailey Levels of Ability | Proposed Measurement points: week 0, 6, 12, 18
  The Chailey Levels of Ability is a scale, which measures motor ability in children and young adults with motor impairment and requires no specialised equipment or environment. It is an observational scale that details physical ability at low levels and can record discrete changes in ability. All participants will be observed in lying postures, including prone and supine where possible, and sitting, with and without support.
Change in Caregiver Priorities & Child Health Index of Life with Disabilities questionnaire | Proposed Measurement points: week 0, 6, 12, 18
  The Caregiver Priorities & Child Health Index of Life with Disabilities consists of 37 items distributed among six sections representing the following domains: (1) Activities of daily living/personal care (2) Positioning, transferring and mobility (3) Comfort and emotions (4) Communication and social interaction (5) Health (6) Overall quality of life. At T0 Baseline, caregivers will complete Section 7, rating the importance of each of the items' contribution to their child's quality of life.
Change in self-reported general health | Proposed Measurement points: serial weekly measurements from week 0-18.
  Participant/caregivers will be asked to report any changes in general health that may be related / unrelated to the study variables.
Change in self-reported change in postural management care plan | Proposed Measurement points: serial weekly measurements from week 0-18.
  Participant/caregivers will be asked to report any pharmaceutical and/or non-pharmaceutical changes in the individual postural management care plan that may be related / unrelated to the study variables.
Change in self-reported change in respiratory management care plan | Proposed Measurement points: serial weekly measurements from week 0-18.
  Participant/caregivers will be asked to report any pharmaceutical and/or non-pharmaceutical changes in the individual respiratory management care plan that may be related / unrelated to the study variables.
Number and category of (Serious) Adverse Events ((S)AE) | Proposed Measurement points: serial weekly measurements from week 0-18.
  Participant/caregivers will be asked to report any "new symptoms" or "worsening symptoms" that may be related / unrelated to the study. This includes action in response to an (S) AE, including primary care consultation (from general practitioner, paediatrician, nurse, therapist etc.), emergency department admission or hospital admission.
Overall Intervention Adherence | Proposed Measurement points: serial weekly measurements from week 6-12.
  Treating therapist will report adherence, recording the number of sessions not attended and reason for non-attendance established via discussion with participant/caregiver during weekly telephone contact.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Marsden, PhD, Study Chair — University of Plymouth
Locations (3):
- United Kingdom (3):
  - Bidwell Brook School, Dartington, Devon
  - John Parkes Unit, Torbay Hospital, Torbay and South Devon NHS Foundation Trust, Torquay, Devon
  - Mayfield School, Torquay

REFERENCES:
- [Background] Morris C, Janssens A, Tomlinson R, Williams J, Logan S. Towards a definition of neurodisability: a Delphi survey. Dev Med Child Neurol. 2013 Dec;55(12):1103-8. doi: 10.1111/dmcn.12218. Epub 2013 Aug 5. PMID 23909744
- [Background] Gibson N, Blackmore AM, Chang AB, Cooper MS, Jaffe A, Kong WR, Langdon K, Moshovis L, Pavleski K, Wilson AC. Prevention and management of respiratory disease in young people with cerebral palsy: consensus statement. Dev Med Child Neurol. 2021 Feb;63(2):172-182. doi: 10.1111/dmcn.14640. Epub 2020 Aug 9. PMID 32803795
- [Background] Winfield NR, Barker NJ, Turner ER, Quin GL. Non-pharmaceutical management of respiratory morbidity in children with severe global developmental delay. Cochrane Database Syst Rev. 2014 Oct 19;2014(10):CD010382. doi: 10.1002/14651858.CD010382.pub2. PMID 25326792
- [Background] Bradley JM, Moran FM, Elborn JS. Evidence for physical therapies (airway clearance and physical training) in cystic fibrosis: an overview of five Cochrane systematic reviews. Respir Med. 2006 Feb;100(2):191-201. doi: 10.1016/j.rmed.2005.11.028. PMID 16412951
- See also: The National Confidential Enquiry into Patient Outcome and Death. Each and Every Need. 2018. London — https://www.ncepod.org.uk/
- See also: Bruce, S. and Stanley, D. Standards of Practice for Physiotherapists Working with adults with a learning disability. 2020 — https://www.csp.org.uk/news/2019-11-19-standards-practice-working-adults-learning-disability-are-launched
- See also: Roberts, D. Bounce Benefits, Physiotherapy Frontline. 2006. 12(3); 12-14. — http://www.csp.org.uk/frontline/article/bounce-benefits